CLINICAL TRIAL: NCT02274883
Title: The Effect of Feeding Infant Formula With Enriched Protein Fractions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Collaborators: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 6027
Record Dates: First submitted 2014-10-16; First posted 2014-10-24 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Cognitive Ability, General

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enriched Protein Fractions (Experimental): This group is given Infant formula with enriched protein fractions.
  Interventions: Dietary Supplement: Enriched Protein Fractions
- Protein Fractions (Active Comparator): This group is given Infant formula with protein fractions.
  Interventions: Dietary Supplement: Protein Fractions

INTERVENTIONS:
Dietary Supplement: Enriched Protein Fractions — Enriched protein fractions
  Arms: Enriched Protein Fractions
Dietary Supplement: Protein Fractions — Protein fractions
  Arms: Protein Fractions

SUMMARY:
This study is intended to evaluate the nutritive effects of study formulas on growth and cognitive outcomes.

DETAILED DESCRIPTION:
To evaluate the nutritive effects of study formulas on growth and cognitive outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 10-14 days of age
* Exclusively formula-fed
* Singleton birth
* Gestational age of 37-42 weeks
* Birth weight of 2500g to 4000g
* Signed Informed Consent Form

Exclusion Criteria:

* History of underlying metabolic or chronic disease
* Congenital malformation
* Condition which is likely to interfere with food ingestion, normal growth, development and evaluation
* Evidence of feeding difficulties or intolerance
* Immunocompromised
* Head/brain disease/injury

Ages: 10 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 451 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Infant cognitive development | At 12 months of age
  Cognitive Scale of Bayley-III is used as the assessment tool.

SECONDARY OUTCOMES:
Infant cognitive development | At 18 months of age
  Cognitive Scale of Bayley-III is used as the assessment tool.
Infant language and motor skills | At 4, 6, 9, 12 and 18 months of age
  Ages and Stages Questionnaire, MacArthur-Bates Communicative Development Index, Language Scale and Motor Scale of Bayley-III are used as the assessment tool.
Infant acquisition of social and emotional milestones and adaptive development | At 4, 6, 9, 12 and 18 months of age
  Ages and Stages Questionnaire, social-emotional scale and adaptive behavior scale of Bayley-III are used as assessment tool.
Infant temperament | At 12 and 18 months of age
  Carey Scale is used as assessment tool.
Infant attention capabilities | At 12 and 18 months of age
  Single Object Attention and Free Play Tasks is used as assessment tool.
Physical development | At 14, 30, 42, 60, 90, 120, 180, 275, 365, and 545 days of age
  Body weight, length and head circumference are measured.
Stool characteristics | At 14, 30, 42, 60, 90, 120, 180, 275 and 365 days of age
  According to the recall of parents during the last 24 hours.
Formula intake | At 30, 42, 60, 90, 120, 180, 275 and 365 days of age
  According to the recall of parents during the last 24 hours.
Fecal microbiome and metabolome profile | Average of 14 days of age and 120 days of age
  Fecal microbiome analysis is done at average of 14 days and 120 days of age. While metabolome profile analysis is done at only average of 120 days of age.
Medically-confirmed Adverse Events | Up to 19 months of age

CONTACTS AND LOCATIONS:
Overall Officials: John Colombo, Doctor, Study Chair — University of Kansas; Fei Li, Doctor, Study Chair — Shanghai Children's Medical Center; Bryan Liu, Doctor, Study Director — Mead Johnson Nutrition
Locations (3):
- China (3):
  - Fuyang Fifth People's Hospital, Fuyang, Anhui
  - Fuyang Maternal and Child Health Institute, Fuyang, Anhui
  - Yinquan Maternal and Child Health Institute, Fuyang, Anhui

REFERENCES:
- [Derived] Chichlowski M, Bokulich N, Harris CL, Wampler JL, Li F, Berseth CL, Rudolph C, Wu SS. Effect of Bovine Milk Fat Globule Membrane and Lactoferrin in Infant Formula on Gut Microbiome and Metabolome at 4 Months of Age. Curr Dev Nutr. 2021 Apr 2;5(5):nzab027. doi: 10.1093/cdn/nzab027. eCollection 2021 May. PMID 33981943
- [Derived] Li F, Wu SS, Berseth CL, Harris CL, Richards JD, Wampler JL, Zhuang W, Cleghorn G, Rudolph CD, Liu B, Shaddy DJ, Colombo J. Improved Neurodevelopmental Outcomes Associated with Bovine Milk Fat Globule Membrane and Lactoferrin in Infant Formula: A Randomized, Controlled Trial. J Pediatr. 2019 Dec;215:24-31.e8. doi: 10.1016/j.jpeds.2019.08.030. Epub 2019 Oct 24. PMID 31668885